CLINICAL TRIAL: NCT00662116
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Evaluate the Effects of Alagebrium on Exercise in Subjects With Diastolic Heart Failure
Brief Title: Beginning a Randomized Evaluation of the AGE Breaker Alagebrium in Diastolic Heart Failure (BREAK-DHF-I)
Acronym: BREAK-DHF-I
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been terminated early due to financial constraints.
Sponsor: Synvista Therapeutics, Inc (Industry)
Responsible Party: Carl Mendel, MD/Chief Medical Officer, Synvista
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-711-0530
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Diastolic Heart Failure
Keywords: diastolic heart failure
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — alagebrium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: alagebrium
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alagebrium — 200 mg (two 100 mg tablets) two times daily for 24 weeks
  Other Names: ALT-711
  Arms: 1
Drug: placebo — placebo tablets - two tablets taken twice daily
  Arms: 2

SUMMARY:
This study is being done to evaluate the safety and effectiveness of alagebrium in subjects diagnosed with diastolic heart failure. The primary assessment for effectiveness is the assessment of exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetes or hypertension requiring therapy
* EF >/= 45% via echo within 1 year and evidence of diastolic heart failure via echo measurement of E/E'>/= 12 determined by echo within 1 year
* previous hospitalization for heart failure or previous BNP >100 pg/mL.

Exclusion Criteria:

* Clinically significant valvular disease
* history of stroke/TIA or reversible ischemic neurological defect w/i 6 mths
* history of acute MI within 6 months
* severe COPD
* active or treated malignancies (except basal cell carcinoma)
* significant systemic illnesses that would prohibit completion of the study or compliance

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy measure will be exercise tolerance as assessed utilizing the 6 Minute Walk Test | Assessed at baseline, week 12 and week 24

SECONDARY OUTCOMES:
QOL as assessed by the Kansas City Cardiomyopathy Questionnaire | baseline, week 12 and week 24
To assess New York Heart Association Classification | Baseline, week 12 and week 24
To evaluate cardiovascular death or hospitalization for heart failure | Will be assessed during the entire 24 wk trial

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Pitt, MD, Principal Investigator — University of Michigan
Locations (30):
- United States (30):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Anaheim, California
  - Bakersfield, California
  - La Jolla, California
  - Roseville, California
  - Jacksonville, Florida
  - Miami, Florida
  - St. Petersburg, Florida
  - Covington, Georgia
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Auburn, Maine
  - South Portland, Maine
  - Ayer, Massachusetts
  - Lincoln, Nebraska
  - Ridgewood, New Jersey
  - Albany, New York
  - Stony Brook, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Fairfield, Ohio
  - Sandusky, Ohio
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Lackland Airforce Base, Texas
  - Milwaukee, Wisconsin